CLINICAL TRIAL: NCT01751295
Title: Effect of Statin on the Post-interventional Coronary Microcirculation Dysfunction
Brief Title: Statin and Post-interventional Coronary Microcirculation Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Ho Choi, professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-08-052
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- atorvastatin (Active Comparator): PCI with atorvastatin pre-treatment group
  Interventions: Drug: Atorvastatin, pre-treatment 80 mg/day for 4 days before PCI
- control (No Intervention): PCI without atorvastatin pre-treatment group

INTERVENTIONS:
Drug: Atorvastatin, pre-treatment 80 mg/day for 4 days before PCI
  Other Names: lipinon
  Arms: atorvastatin

SUMMARY:
The purpose of this study is to evaluate the effect of statin on the coronary microcirculation dysfunction measured after percutaneous coronary intervention.

DETAILED DESCRIPTION:
Development of peri-procedural myocardial infarction following percutaneous coronary intervention (PCI) is not uncommon and affects long-term prognosis. Clinical studies have shown that pre-treatment with atorvastatin reduced peri-procedural myocardial infarction in patients with stable angina. The mechanism of peri-procedural myocardial infarction is presumed to be microvascular embolization. However the direct causal relationship between statin pretreatment and prevention of microvascular dysfunction has not been investigated yet.

In this study, we will recruit symptomatic angina patients who have clinical indication of coronary angiography. At the time of enrollment, patients will be randomly assigned to pre-treatment group (atorvastatin 80 mg/d for 4 days) or control group. Percutaneous coronary intervention (PCI) will be perfomed based on the result of diagnostic coronary angiography by decision of attending physician. When PCI is performed, fractional flow reserve (FFR) and index of microvascular resistance (IMR) will be measured before and after the procedure. Periprocedural myocardial infarction will be defined by post-PCI cardiac biomarker. All patients will be followed for adverse cardiac events for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* A. Finished informed consent
* B. Stable angina with clinical indication of coronary angiography
* C. Age ≥ 21 year and ≤ 80 year

Exclusion Criteria:

* A.Without informed consent
* B.PCI target lesion is not adequate or not indicated for FFR/IMR study
* C.Prior myocardial infarction or interventional procedure for PCI target vessel
* D.Myocardial infarction within 30 days
* E.Usage of statin, current or within 1 month
* F.Prior bypass surgery
* G.Impaired renal function (Creatinine > 2.0 mg/dL)
* H.Impaired left ventricular function (ejection fraction < 40%)
* I.Active hepatitis or abnormal hepatic transaminase level (> 3 ULN)
* J.Contraindication for long-term antiplatelet agent or statin
* K.Planning or potential of pregnancy
* L.Neoplastic disease without evidence of treatment completion
* M.Impaired general condition

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Post-procedural IMR of PCI target vessel Post-procedural IMR of PCI target vessel | within 1 year after PCI

SECONDARY OUTCOMES:
Post-procedural troponin I | within 1 year after PCI
Post-procedural FFR | within 1 year after PCI
Post-procedural IMR comparison of target vessel with non-target vessel | within 1 year after PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gang nam-Gu, Ilwon-Dong, South Korea